CLINICAL TRIAL: NCT01805661
Title: Assessment of Early Ambulation and Participation in Rehabilitation Program in Patients Receiving Continuous Adductor Canal Block With Ultrasound Guided Posterior Capsular Knee Injection vs Continuous Femoral Nerve Block With Tibial Nerve Block Following Total Knee Replacement.
Brief Title: Adductor Canal Block With Posterior Capsular Injection for Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-10-002
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Osteoarthritis
Keywords: early ambulation; knee arthroplasty
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral With Tibial Nerve Block (Active Comparator): Continuous femoral nerve block with catheter and selective tibial nerve block in the popliteal fossa
  Interventions: Procedure: Femoral with Tibial Nerve Block
- Canal Block and Capsular Injection (Experimental): Adductor canal block with a continuous catheter and ultrasound guided posterior capsular injection with local anesthetic solution.
  Interventions: Procedure: Canal Block and Capsular Injection

INTERVENTIONS:
Procedure: Canal Block and Capsular Injection — Continuous Adductor canal block with 15-30ml of ropivacaine 0.1% with epinephrine 1:400,000 followed by an infusion of ropivacaine 0.1% at 6 ml per hour for 2 days post operatively. This is combined with ultrasound guided posterior capsular knee injection with 30 ml ropivacaine 0.1% with epinephrine 1:400,000.
  Arms: Canal Block and Capsular Injection
Procedure: Femoral with Tibial Nerve Block — Continuous femoral nerve block with 15 ml of ropivacaine 0.1% followed by an infusion of ropivacaine 0.1% at 6 ml per hour for 2 days after surgery combined with tibial nerve block in the popliteal fossa with ropivacaine 0.1% up to 15 ml.
  Arms: Femoral With Tibial Nerve Block

SUMMARY:
To compare early ambulation and ability to participate in rehabilitation in patients undergoing total knee replacement using two different nerve block techniques for pain control. The 2 methods are 1) Adductor canal block with posterior capsular injection 2) femoral nerve block with tibial nerve block

DETAILED DESCRIPTION:
Early mobilization in the postoperative period is important to the success of surgery following total knee replacement. However, severe post-operative pain is an impediment to early implementation of rehabilitaion program. The use of femoral nerve block combined with tibial nerve block as part of a multimodal analgesic program provides effective pain control but causes weakness of the operative extremity preventing patients from bearing weight, exercising the leg and increasing the risk of falls thereby delaying early participation in rehabilitation. Adductor canal block is a new technique that has been described to provide pain control after total knee arthroplasty (1). The advantages of this block is that it could potentially minimize lower extremity weakness because the target nerve (saphenous nerve) blocked in this technique is a purely sensory nerve and does not provide any motor innervation to any muscle groups. Adductor canal block lends itself easily to providing prolonged analgesia because a perineural catheter can be inserted and the block maintained by a continuous infusion of dilute local anesthetic solution for days. A disadvantage of this method is that it may not provide adequate analgesia for posterior knee pain in the early postoperative period. By combining adductor canal block with ultrasound guided posterior and antero-medial knee injection, the posterior knee pain can be controlled effectively. Posterior and antero-medial knee injection of local anesthetic solution has been used as a method of controlling posterior knee pain after total knee arthroplasty (2).

ELIGIBILITY:
Inclusion Criteria:

* Patients having primary, unilateral total knee arthroplasty
* ages 18 - 80

Exclusion Criteria:

* history of neurological disease
* neuropathy
* diabetes
* major systemic illness
* pregnancy
* chronic narcotic use
* allergy to local anesthetic solution or NSAIDS
* inability to give consent or cooperate with the study protocol
* BMI> 40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ability to ambulate post operatively. | Up to 3 days (72 hours) post surgery.
  Ability to ambulate and perform tasks of the rehabilitation program and reach rehabilitation milestones after total knee arthroplasty.

SECONDARY OUTCOMES:
Pain scores at rest and with knee flexion. | Up to 3 days ( 72 hours) after surgery
  Measures of pain score using numeric pain rating scale (0=no pain, 10=worst pain) completed by patient in recovery room and every 6 hours for a 72 hour period after discharge from recovery room.
Pain Medication Consumption | Up to 3 days (72 hours) post surgery
  Amount of opioid consumption post surgery for 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, M.D., Principal Investigator — Saint Francis Hospital and Medical Center
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States